CLINICAL TRIAL: NCT01617135
Title: A Randomized, Placebo-Controlled, Phase 2 Study of the Safety, Pharmacokinetics and Pharmacodynamics of CVT-310 (Levodopa Inhalation Powder) in Patients With Parkinson's Disease and Motor Response Fluctuations ("Off Episodes")
Brief Title: Safety, Pharmacokinetics and Efficacy Study of CVT-301 Inpatients With Parkinson's Disease and "Off" Episodes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Acorda Therapeutics (Industry)
Collaborators: Michael J. Fox Foundation for Parkinson's Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CVT-301-002; 2012-000181-37 (EudraCT Number)
Record Dates: First submitted 2012-05-07; First posted 2012-06-12 (Estimated); Last update posted 2017-07-27 (Actual); Status verified 2017-07

CONDITIONS: Idiopathic Parkinson's Disease
Keywords: Parkinson's disease; Motor fluctuations; levodopa; inhaled drugs; Motor fluctuation ("off episodes")
MeSH Terms: conditions — Parkinson Disease | interventions — carbidopa, levodopa drug combination; Carbidopa; Levodopa

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- CVT-301 Low Dose (Experimental): CVT-Low; levodopa inhalation powder (LIP)
  Interventions: Drug: CVT-301
- CVT-301 High Dose (Experimental): CVT-High; levodopa inhalation powder (LIP)
  Interventions: Drug: CVT-301
- Inhaled Placebo (Placebo Comparator): Inhaled placebo powder
  Interventions: Drug: Placebo
- Oral Sinemet (carbidopa/levodopa) (Active Comparator): Open-label oral carbidopa/levodopa (CD/LD)
  Interventions: Drug: Sinemet (carbidopa/levodopa)

INTERVENTIONS:
Drug: CVT-301
  Arms: CVT-301 Low Dose
Drug: Placebo
  Arms: Inhaled Placebo
Drug: Sinemet (carbidopa/levodopa)
  Arms: Oral Sinemet (carbidopa/levodopa)
Drug: CVT-301
  Arms: CVT-301 High Dose

SUMMARY:
The purpose of this study is to determine the safety, efficacy and pharmacokinetics following administration of CVT-301 in treatment of "off" episodes in Parkinson's Disease patients.

DETAILED DESCRIPTION:
Treatment options for patients with motor response fluctuations are limited. Most commonly, "off" episodes are managed by adjusting the dose interval of their standard oral medications or by self-administration of unscheduled doses of oral Parkinson's medication. Due to the variability in levodopa absorption following oral dosing, resumption of motor function is unreliable and may be delayed for an hour or more. CVT-301 delivers levodopa using a simple inhaler, resulting in rapid increases in levodopa blood levels and is expected to result in rapid restoration in motor function for patients experiencing "off" episodes.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic Parkinson's Disease (PD) diagnosed between the ages of 30 and 80 years;
* Hoehn and Yahr Stage 1-3 in an "on" state;
* Require levodopa-containing medication regimen at least 4 times during the waking day;
* Experience motor fluctuations with a minimum of 2 hours of average daily "off" time per waking day (excluding early morning "off" time) and demonstrate levodopa responsiveness;
* Are on stable PD medication regimen.

Exclusion Criteria:

* Pregnant or lactating females;
* Previous surgery for PD or plan to have stereotactic surgery during the study period;
* History of psychotic symptoms requiring treatment, or suicide ideation or attempt within last year;
* Adequate lung function as measured by spirometry;
* Any significant condition, severe concurrent disease, abnormality or finding that would make patients unsuitable or may compromise patient safety.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2012-05; Primary Completion 2012-11 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Safety | change from baseline up to 13 weeks
  Adverse experiences, ECGs, clinical laboratory evaluation, pulmonary function

SECONDARY OUTCOMES:
Pharmacodynamics | 3 hours post-dose
  Time to onset of meaningful "on" and "off" states (patient- and examiner-assessed) UPDRS III motor score Tapping test Dyskinesia
Pharmacokinetics | 3 hours post-dose
  Serial blood draw for determination of plasma concentration-time profile

CONTACTS AND LOCATIONS:
Locations (7):
- Israel (2):
  - Civitas Clinical Site #6, Petah Tikva
  - Civitas Clinical Site #5, Tel Aviv
- Serbia (2):
  - Civitas Clinical Site #4, Belgrade
  - Civitas Clinical Site #7, Belgrade
- United Kingdom (3):
  - Civitas Clinical Site #1, Glasgow
  - Civitas Clinical Site #3, Newcastle
  - Civitas Clinical Site #2, Norwich

REFERENCES:
- See also: Related Info — https://foxtrialfinder.michaeljfox.org/